CLINICAL TRIAL: NCT03494881
Title: Mepolizumab for the Treatment of Chronic Spontaneous Urticaria: An Open-label, Single-arm, Exploratory Study
Brief Title: Mepolizumab for the Treatment of Chronic Spontaneous Urticaria
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jason Sluzevich MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-009322
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Mepolizumab for the treatment of chronic spontaneous urticaria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): This is an open-label pilot investigation and all study participants are assigned to active treatment. There is no placebo arm in this study.
  Interventions: Drug: Nucala

INTERVENTIONS:
Drug: Nucala — All study participants will receive Nucala (2) 100mg SQ injections administered at two different anatomical sites at week zero, 2,4,6, and 8 for a total of 5 doses.
  Other Names: Mepolizumab

SUMMARY:
This is an exploratory study designed to generate preliminary data in evaluating the efficacy of Nucala in the treatment of chronic spontaneous urticaria.

DETAILED DESCRIPTION:
This is an open-label, single arm exploratory study of mepolizumab in the treatment of CSU. The primary endpoint will be the mean reduction in the seven day urticaria activity score (UAS7) before and after 10 weeks of treatment with mepolizumab. Secondary endpoints will be the mean reduction of the urticaria control test (UCT) score and the weekly itch severity score (ISS) before and after treatment. Enrollment examination will include a standardized history and examination, baseline UCT score, CBC with differential, serum IgE level, chronic urticaria index, IgE Fc receptor antibody functional assay, and a 4 mm punch biopsy of lesional skin to confirm the urticarial tissue reaction includes eosinophils and is not neutrophilic predominant. Patients will discontinue all anti-histamines and start cetirizine 10 mg PO BID which may be continued throughout the study duration. Patients will be provided with a log book to track daily urticaria signs and symptoms in a standardized manner for UAS scoring. At week 0 (enrollment visit +7 days), baseline UAS7 and ISS score will be assessed and skin biopsy results reviewed. Patients with a confirmatory skin biopsy will receive 200 mg SC of mepolizumab at week 0,2,4,6,and 8. UAS-7 and weekly ISS score will be calculated at week 0, 4, 8, and 10. UCT scoring will be calculated at week 0 and at week 10. Repeat CBC with differential, serum IgE level, and measures of basophil serum activation (chronic urticaria index, IgE FC Receptor antibody functional assay) will be assessed at week 10. Attached to this document is a protocol summary.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older.
* Clinical and/or histopathological diagnosis of conventional CSU
* Unresponsive to oral antihistamine therapy
* Good general health as confirmed by medical history
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion Criteria:

* Vulnerable study population
* If you are female and pregnant
* Biopsy proven neutrophilic rich urticaria
* Known history of adverse reaction to mepolizumab (Nucala)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2025-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Sluzevich, M.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: This was an open-label pilot investigation and all study participants were assigned to active treatment. There was no placebo arm in this study.
  Nucala: All study participants received Nucala (2) 100mg SQ injections administered at two different anatomical sites at week zero, 2,4,6, and 8 for a total of 5 doses.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Urticaria Activity Score (UAS7)
Description: Study participants documented their chronic spontaneous urticaria (CSU) symptoms using a diary, daily scoring for a) the number of wheals [none (=0 points), <10 (=1 point), 10-50 (=2 points), or >50 per day (=3 points)], and b) the intensity of pruritus [none (=0 points), mild (=1 point), moderate (=2 points), severe (=3 points)]. The daily UAS score is summed over a week to calculate the UAS7 score (range: 0-42). Participants were considered responders if they had ≥ 95% reduction in baseline UAS7 score and non-responders if they had <95% reduction in baseline UAS7 score.
Time Frame: Baseline to 10 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  Responders | 3
  Non-Responders | 7

2. Secondary Outcome: Change in Short Form Urticaria Control Test Score (S-UCT)
Description: The short form urticaria control test (S-UCT) is a more recently developed and validated outcome instrument to retrospectively assess urticaria control. The S-UCT consists of 4 questions with each question having 5 answer options scored 0-4 with low points indicating high disease activity and low disease control. The minimum and maximum S-UCT scores are 0-16 with 16 points indicating complete disease control. Participants were considered responders if they had ≥ 95% reduction in baseline S-UCT score and non-responders if they had <95% reduction in baseline S-UCT score.
Time Frame: Baseline to 10 weeks
Population: 10 total participants were analyzed. Those 10 participants were further broken down into the following categories non-responders (7) and responders (3), respectively.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
score on a scale
  Responders: number analyzed (Participants) | 3
  Responders | 12.3 [0 to 16]
  Non-responders: number analyzed (Participants) | 7
  Non-responders | 0.71 [0 to 16]

3. Secondary Outcome: Change in Long Form Urticaria Control Test (L-UCT) Score
Description: The long form urticaria control test (L-UCT) is a more recently developed and validated outcome instrument to retrospectively assess urticaria control. The L-UCT consists of 8 questions with each question having 5 answer options scored 0-4 with low points indicating high disease activity and low disease control. The minimum and maximum L-UCT scores are 0-32 with 32 points indicating complete disease control. Participants were considered responders if they had ≥ 95% reduction in baseline L-UCT score and non-responders if they had <95% reduction in baseline L-UCT score.
Time Frame: Baseline to 10 Weeks
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
score on a scale
  Responders: number analyzed (Participants) | 3
  Responders | 21.3 [0 to 32]
  Non-Responders: number analyzed (Participants) | 7
  Non-Responders | 1.6 [0 to 32]

4. Secondary Outcome: Change in Itch Severity Score (ISS)
Description: The weekly itch severity score measures the intensity and impact of itching (pruritus). It is calculated using the pruritus score of the daily Urticaria Activity Score (UAS) score summed over a week. Scores range from 0 to 21 with higher scores indicating worse itching. Participants were considered responders if they had ≥ 95% reduction in baseline ISS score and non-responders if they had <95% reduction in baseline ISS score.
Time Frame: Baseline to 10 weeks
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
score on a scale
  Responders: number analyzed (Participants) | 3
  Responders | 13 [0 to 21]
  Non-Responders: number analyzed (Participants) | 7
  Non-Responders | 1 [0 to 21]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through end of study participation, approximately 10 weeks.
Description: This study defined an adverse event as an untoward or undesirable experience associated with the use of Mepolizumab (Nucala) in a research subject. Adverse events were collected through non-directed questioning of subjects at each follow-up visit.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=10)
Facial Swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03494881/Prot_SAP_000.pdf